CLINICAL TRIAL: NCT00689039
Title: A Two-part, Single-centre, Open (Part A) Single Blind (Part B), Randomised, Placebo-controlled Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics After Single Doses With and Without Food and Multiple Ascending Oral Doses of AZD1305 Extended-release Tablet in Healthy & Elderly Subj
Brief Title: Study of an Extended Release (ER) Tablet, Single and Repeated Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3190C00004; 2006-006356-35 (EudraCT No)
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: AZD1305; safety; pharmacokinetics; multiple ascending doses; Safety and pharmacokinetics
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD1305 ER tablet
  Interventions: Drug: AZD1305
- B (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — ER tablet, administered as single and repeated doses.
  Arms: A
Drug: Placebo — Tablet, administered as single and repeated doses.
  Arms: B

SUMMARY:
The purpose is to study the safety and tolerability of increasing doses of AZD1305 and how the medication is metabolised by the body (how it is taken up, distributed, and how it disappears from the body). The study is performed in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI=weight/height2) of 19 to 27 kg/m2
* Clinically normal physical findings, laboratory values and resting ECG as judged by the investigator

Exclusion Criteria:

* ECG findings outside normal range
* Potassium outside normal reference values

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Adverse events, ECG, vital signs, physical examination, laboratory variables, body temperature and weight | During the study

SECONDARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Marianne Hartford, MD, PhD, Principal Investigator — AstraZeneca, Clinical Pharmacology Unit at Sahlgrenska University Hospital, Sweden
Locations (1):
- Research Site, Gothenburg, Sweden